CLINICAL TRIAL: NCT03976206
Title: Autologous Very Small Embryonic-like Stem Cells(VSELs) for Facial Skin Antiaging
Brief Title: Very Small Embryonic-like Stem Cells for Facial Skin Antiaging
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Policy changes have contributed to the failure to carry out smoothly
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Guangzhou Four-Leaf Clover HealthTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSEL-face
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-06

CONDITIONS: Stem Cell Transplant Complications; Skin Inflammation
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Intervention Model Description: In the experimental group, VSELs will be injected in left preauricular area of every volunteer, followed by skin pathology to compare the improvement of skin aging with the skin of right preauricular area. In the control group, platelet-rich plasma will be injected to the left preauricular area of every volunteer.
Who Masked: Investigator
Masking Description: The volunteers will be randomly arranged to enter the experimental group or the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VSEL Max (Experimental): We carried out the subdermal application of VSELs with a 1-mL syringe (90,000 cells in 0.4 mL plate-rich plasma) coupled to a 30-gauge needle, in the left preauricular area (1-cm2 area), 2 cm distal from the tragus
  Interventions: Biological: Very small embryonic-like stem cell
- VSEL Medium (Experimental): We carried out the subdermal application of VSELs with a 1-mL syringe (60,000 cells in 0.4 mL plate-rich plasma) coupled to a 30-gauge needle, in the left preauricular area (1-cm2 area), 2 cm distal from the tragus
  Interventions: Biological: Very small embryonic-like stem cell
- VSEL Mini (Experimental): We carried out the subdermal application of VSELs with a 1-mL syringe (30,000 cells in 0.4 mL plate-rich plasma) coupled to a 30-gauge needle, in the left preauricular area (1-cm2 area), 2 cm distal from the tragus
  Interventions: Biological: Very small embryonic-like stem cell
- Control (No Intervention): Subcutaneous injection of 0.4 mL platelet-rich plasma in the same part of the experimental group

INTERVENTIONS:
Biological: Very small embryonic-like stem cell — We carried out the subdermal application of VSELs with a 1-mL syringe (volume, 0.4 mL) coupled to a 30-gauge needle, in the left preauricular area (1-cm2 area), 2 cm distal from the tragus
  Other Names: VSEL
  Arms: VSEL Max; VSEL Medium; VSEL Mini

SUMMARY:
The aim of this study is the safety and efficacy of autologous very small embryonic-like stem cells(VSELs) to facial skin antiaging.

DETAILED DESCRIPTION:
VSELs come from the patient's peripheral blood, and will be injected in left preauricular area, followed by skin pathology to compare the improvement of skin aging. Two 0.5 × 1 cm fragments of skin and subcutaneous tissue was removed from bilateral preauricular areas for morphologic analysis by optical and electron microscopy. Histologic analysis of skin biopsy specimens was performed by hematoxylin and eosin, picrosirius red (for visualization of collagen), and orcein (for visualization of elastic fibers) staining.

ELIGIBILITY:
Inclusion Criteria:

• Healthy volunteers with anti-aging willingness

Exclusion Criteria:

* Metabolic and systemic diseases such as diabetes and atherosclerosis
* Facial skin diseases such as herpes, eczema, skin rash, systemic lupus erythematosus, dermatomyositis, connective tissue disease
* Endocrine disorders and cancer patients Blood disease patients, thrombocytopenia or dysfunction, hypofibrinemia or anticoagulant therapy, long-term use of aspirin

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 1 week
  Swelling in the skin at the injection site
Incidence of treatment-emergent adverse events | 1 week
  Color change, pain in the skin at the injection site
Incidence of treatment-emergent adverse events | 1 week
  Pain in the skin at the injection site

SECONDARY OUTCOMES:
Short-term changes in skin histopathology | 3-6 months after injection
  Two 0.5 × 1 cm fragments of skin and subcutaneous tissue was removed from the bilateral preauricular areas for morphologic analysis by optical and electron microscopy
Long-term changes in skin histopathology | 12 months after final injection
  Two 0.5 × 1 cm fragments of skin and subcutaneous tissue was removed from the bilateral preauricular areas for morphologic analysis by optical and electron microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No